CLINICAL TRIAL: NCT06246552
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Single-dose Phase 2 Study of the Safety and Efficacy of JTM201 (Botulinum Toxin Type A) to Treat Moderate or Severe Glabellar Lines
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of JTM201 to Treat Moderate or Severe Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jetema USA Inc. (Industry)
Responsible Party: Sponsor
Organization: Jetema Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: J-001-US
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JTM201 (Experimental): Botulinum toxin
  Interventions: Biological: JTM201
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JTM201 — JTM201 20U in 0.5mL
  : JTM201 will be injected via IM in 5 glabellar location 0.1mL (4U / 0.1mL) at each location
  Arms: JTM201
Biological: Placebo — Placebo 20U in 0.5mL
  : Placebo will be injected via IM in 5 glabellar location 0.1mL (4U / 0.1mL) at each location
  Arms: Placebo

SUMMARY:
This is Multicenter, Randomized, Double-blind, Placebo-controlled, Single-dose Study to evaluate Safety and Efficacy of JTM201 in patients with Moderate or Severe Glabellar Lines

DETAILED DESCRIPTION:
This is Multicenter, Randomized, Double-blind, Placebo-controlled, Single-dose Study to evaluate Safety and Efficacy of JTM201 in patients with Moderate or Severe Glabellar Lines. Treatment period is 180 days and evaluation of the safety is the primary endpoint

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age based on the date of the written informed consent form.
* Subject is able to provide written informed consent and comply with study procedures.
* Subject has moderate or severe glabellar lines on maximum frown as assessed by the investigator and subject using the GLS (score of 2 or 3).

Exclusion Criteria:

* Previous insertion of permanent material in the glabellar area including the forehead.
* Planned treatment with botulinum toxin of any serotype in any other body region during the study period.
* Pregnant or breastfeeding (directly or via pump); or planning to become pregnant during the study.
* Known allergy or hypersensitivity to botulinum toxin or product excipients.
* Participation in another interventional clinical study ≤30 days of Visit 1: Screening.
* Planning to donate, bank, or retrieve eggs (ova, oocytes) or donate sperm during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
TEAE | 180 days
  Treatment-emergent AEs (TEAEs) from Baseline through end of followup
SAE | 180 days
  Serious AEs (SAEs) from the screening period through end of follow-up

OTHER OUTCOMES:
Glabellar Line Scale (GLS) | 30 days
  Proportion of subjects who achieve a ≥ 2-point improvement in GLS at maximum frown by IA and SSA from Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No